CLINICAL TRIAL: NCT05379205
Title: Multidisciplinary Prehabilitation and Postoperative Rehabilitation for Avoiding Complications in Patients Undergoing Resection of Colon Cancer: ONCOFIT Study
Brief Title: Multidisciplinary Prehabilitation and Postoperative Rehabilitation in Patients Undergoing Resection of Colon Cancer
Acronym: ONCOFIT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: Hospital Clinico Universitario San Cecilio (Other); Universidad de Córdoba (Other)
Responsible Party: Principal Investigator, Francisco Jose Amaro-Gahete, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019529142937
Record Dates: First submitted 2022-04-23; First posted 2022-05-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Colon Cancer; Postoperative Complications
Keywords: Post-surgery complications; Multidisciplinary intervention; Exercise; Dietary behaviour; Psychological support
MeSH Terms: conditions — Colonic Neoplasms; Postoperative Complications; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care/Control Group (Active Comparator): Usual care group will follow the usual institutional pre-surgery care..
  Interventions: Other: Usual Care
- Prehabilitation + Postoperative Programs (PPP) Group (Experimental): PPP group will include 3 complementary modules: (i) supervised physical exercise, (ii) dietary behavior change, and (iii) psychological support.
  Interventions: Behavioral: Prehabilitation program (4 week before the surgery); Behavioral: Postoperative program (12 week after the surgery)

INTERVENTIONS:
Behavioral: Prehabilitation program (4 week before the surgery) — This intervention will include 3 complementary modules: (i) supervised physical exercise: aerobic and strength High Intensity Interval Training (HIIT), 3 times per week (ii) dietary behavior change: nutritional talk + an informative brochure + a video summary, a session per week and (iii) psychological support: psychoeducation, written and verbal emotional expression, promotion of coping strategies, progressive muscle relaxation training, problem-solving and social skills, and self-efficacy enhancing, among others. This psychological component will also include counseling regarding smoking and alcohol cessation and sleep hygiene.
  Arms: Prehabilitation + Postoperative Programs (PPP) Group
Behavioral: Postoperative program (12 week after the surgery) — This intervention will include 3 complementary modules: (i) supervised physical exercise: aerobic and strength High Intensity Interval Training (HIIT), 3 times per week (ii) dietary behavior change: nutritional talk + an informative brochure + a video summary, a session per week and (iii) psychological support: psychoeducation, written and verbal emotional expression, promotion of coping strategies, progressive muscle relaxation training, problem-solving and social skills, and self-efficacy enhancing, among others. This psychological component will also include counseling regarding smoking and alcohol cessation and sleep hygiene.
  NOTE: Both preoperative and postoperative programs will be administer to the participants assigned to the intervention group.
  Arms: Prehabilitation + Postoperative Programs (PPP) Group
Other: Usual Care — Usual care group will follow the usual institutional pre-surgery care: (i) medication management, (ii) assessment of the surgery-derived risks, (iii) smoking cessation and peri-operative blood management. A trained nutritionist will evaluate the nutritional status of all patients at the baseline providing oral protein/vitamin supplementation, when necessary. Patients allocated to the control group will receive basic expert' advice on lifestyle changes.
  Arms: Usual Care/Control Group

SUMMARY:
ONCOFIT is a randomized clinical trial with a two-arm parallel design aimed at determining the influence of a multidisciplinary prehabilitation + postoperative program on post-surgery complications in patients undergoing resection of colon cancer. This intervention will include supervised physical exercise, dietary behavior change, and psychological support comparing its influence to the standard care.

DETAILED DESCRIPTION:
Nowadays, colon cancer is one of the most common types of tumors worldwide being surgical resection the elective therapy for its curation. However, a surgery is a stressful procedure that may involve several postoperative complications. Risk factors for such undesirable events are closely related to lifestyle issues including decreased physical activity levels or dietary unhealthy habits. Recent studies have suggested that the implementation of multidisciplinary prehabilitation and postoperative interventions based on lifestyle habits may be a potential strategy for accelerate post-surgical recovery. To the best of our knowledge, the combined effect of a Prehabilitation + Postoperative Programs (PPP) on post-surgery complications and functional capacity of patients undergoing resection of colon cancer remains unclear. ONCOFIT is a randomized clinical trial with a two-arm parallel design aimed at determining the influence of a multidisciplinary PPP on post-surgery complications in patients undergoing resection of colon cancer. This intervention will include supervised physical exercise, dietary behavior change, and psychological support comparing its influence to the standard care. Primary and secondary endpoints will be assessed at baseline, at preoperative conditions, at the end of the PPP intervention and 1-year post-surgery, including: post-surgery complications, prolonged hospital length of stay, readmissions and emergency department call, functional capacity, patient' reported outcome measures targeted, anthropometry and body composition, clinical markers, physical activity levels and sedentariness, dietary habits, others unhealthy habits, sleep quality and fecal microbiota diversity and composition. Considering the feasibility of the present intervention in a real-life scenario, ONCOFIT will contribute to the standardization of a cost-effective strategy for preventing and improving health-related consequences in patients undergoing resection of colon cancer with an important clinical and economic impact, not only in the scientific community but also in the clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 40 years
* Diagnostic of nonmetastatic colon cancer (i.e., including right, transverse, left, sigmoid, subtotal, total, and hemicolectomy)
* Not participating in a nutritional/ dietary intervention
* Being physical inactive (i.e., not to be participating in any physical exercise program in the last 3 months, or performing less than 600 metabolic equivalents (METS)/week of moderate-vigorous physical activity).
* To be capable and willing to provide informed consent
* Not to suffer from any specific condition that may impede testing of the study hypothesis or make it unsafe to engage in the multidisciplinary intervention (i.e., determined by the research staff).

Exclusion Criteria:

* Medical contraindication for being engaged in an exercise or dietary program.
* Additional surgery planned within the 3-month intervention
* History of another primary invasive cancer
* Planning to receive adjuvant chemotherapy
* To be pregnant
* To present any of the following cardiac conditions: (i) myocardial infarction or coronary revascularization procedure within prior 3 months, (ii) uncontrolled hypertension (i.e., systolic ≥180 mmHg or diastolic ≥100 mmHg), (iii) uncontrolled arrhythmias (iv) valvular disease clinically significant, (v) decompensated heart failure or (vi) to suffer from known aortic aneurysm.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Post-surgery complications | 30-days and 3-months post-surgery
  Post-surgery complications determined by the Comprehensive Complication Index (CCI). Minimum value: 0 // Maximum value: 100. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Post-surgery complications | 1-year post-surgery (i.e., week 57)
  Post-surgery complications determined by the Comprehensive Complication Index (CCI). Minimum value: 0 // Maximum value: 100. Higher scores mean a worse outcome.
Additional surgery-derived events | 1-year post-surgery (i.e., week 57).
  Electronic medical records will be used to register data regarding primary and total prolonged hospital length of stay.
Post-surgery complications | 30-days, 3-months and 1-year post-surgery
  Post-surgery complications determined by the number of patients experiencing complications.
Additional surgery-derived events | 30-days, 3-months and 1-year post-surgery
  Electronic medical records will be used to register data regarding readmissions.
Additional surgery-derived events | 30-days, 3-months and 1-year post-surgery
  Electronic medical records will be used to register data regarding emergency department appointments.
Additional surgery outcomes | 24 hours, 48 hours and 72 hours after the surgical procedure.
  Quality of Recovery Short-form questionnaire (QOR-15). Minimum value: 0// Maximum value: 150. Higher scores mean a better outcome.
  Visual Analogue Scale for abdominal pain. Minimum value: 0 // Maximum value: 100. Higher score mean a worse outcome
Cardiorespiratory fitness | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  Cardiorespiratory fitness measured by the 6-minute walking test (6MWT) distance, expresed in total m.
Upper Limb muscular strength | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  Muscular strength assessed by handgrip strength. Handgrip strength will be determined using a digital hand dynamometer and expressed as total kg.
Lower limb muscular strength | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  Muscular strength assessed by the 30 seconds sit-to-stand test.
Lower limb muscular strenght | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  Muscular strength assessed by the 5 times sit-to-stand test, assessing the time needed to rise 5 times from a seated position without using arms.
Gait speed | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  The 4-meter usual walking speed test will be used to assess the Gait Speed
Health-related quality of life | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  The European Organisation for Research and Treatment of Cancer quality of life questionnaire for patients with colorectal cancer (EORT-QLQ-CR29).
Self-scored depression inventory | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  The Beck Depression Inventory-II questionnaire. Minimum value: 0 // Maximum value: 63. Higher scores mean a worse outcome.
Trait and state anxiety | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  The State-Trait Anxiety Inventory (STAI). Minimum value: 20 // Maximum value: 80. Higher scores mean a worse outcome.
Anxiety and Depression Levels | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  The Hospital Anxiety and Depression Scale (HADS). Minimum value: 0 // Maximum value: 21. Higher scores mean a better outcome.
Mental Adjustment to Cancer | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  The Mini-Mental Adjustment to Cancer. Five sub-scales are measured by this questionnaire: hopeless, anxious preoccupation, fighting spirit, fatalism and cognitive avoidance.
Weight | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  Weight measured with a scale (kg).
Height | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  Height measured with a stadiometer (cm).
Neck, waist and hip circumferences | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  Neck, waist and hip circumferences will be assessed with an anthropometric tape measure (cm).
Bone mineral density | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  Body composition assessment will be obtained through a full-body dual energy X-ray absorptiometry scanner. Bone mineral density in g/cm2.
Lean mass | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  Body composition assessment will be obtained through a full-body dual energy X-ray absorptiometry scanner. Lean mass in kg.
Fat mass | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  Body composition assessment will be obtained through a full-body dual energy X-ray absorptiometry scanner. Fat mass in kg.
Visceral adipose tissue | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  Body composition assessment will be obtained through a full-body dual energy X-ray absorptiometry scanner. Visceral adipose tissue in kg.
Glycemic profile | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  Blood samples will be drawn from patient' antecubital vein in a supine position during the morning after an overnight fasting to assess the glycemic profile. We will obtain plasma glucose (mg/dL) and insulin (mg/dL) levels.
Lipid profile | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  Blood samples will be drawn from patient' antecubital vein in a supine position during the morning after an overnight fasting to assess the lipid profile.
Hepatic transaminases | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  Blood samples will be drawn from patient' antecubital vein in a supine position during the morning after an overnight fasting to assess the hepatic transaminases levels.
Red cells | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  Blood samples will be drawn from patient' antecubital vein in a supine position during the morning after an overnight fasting to assess the red cells levels.
Immunological blood profiles | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  Blood samples will be drawn from patient' antecubital vein in a supine position during the morning after an overnight fasting to assess the immunological blood profiles. The following parameters will be obtained: Leukocytes (10*3 uL), Neutrophils (10*3 uL), Lymphocytes (10*3 uL), Monocytes (10*3 uL), Eosinophils (10*3 uL), Basophils (10*3 uL) and LUC cells (10*3 uL).
Inflammatory factors | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  Blood samples will be drawn from patient' antecubital vein in a supine position during the morning after an overnight fasting to assess the inflammatory factors levels (PCR, leptin, adiponectin, resistin, IL 6, IL 10 and PAI 1; all of them expressed as pg/mL)
Renal function parameters | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  Blood samples will be drawn from patient' antecubital vein in a supine position during the morning after an overnight fasting to assess the renal function parameters (creatinine and urea; both will be expressed in mg/dL)
Tumour markers | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  Blood samples will be drawn from patient' antecubital vein in a supine position during the morning after an overnight fasting to assess the tumour markers levels (CA 19-9, CA 242, CA 72-4, TPA and TPS; all will be expressed as pg/mL))
Hormones | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  Blood samples will be drawn from patient' antecubital vein in a supine position during the morning after an overnight fasting to assess the hormones levels (T3, T4, testosterone, cortisol, estrogens and DHEAs; all will be expressed as pg/mL))
Blood pressure | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  The investigators will also asses systolic and diastolic blood pressure in the right arm at rest.
HOMA index | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  The investigators will calculate the homeostatic model assessment of insulin resistance index (HOMA). HOMA index was calculated as follows: (fasting glucose(mg/dl) x fasting serum insulin (μU/mL))/405.
FLI index | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  The investigators will calculate the fatty liver index (FLI) as a validated surrogate marker of non-alcoholic fatty liver disease.
Cardiometabolic risk | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  The investigators will calculate a cardiometabolic risk score based on the International Diabetes Federation (IDF) criteria. The cardiometabolic risk score is a continuous variable with a mean of 0 and a standard deviation of 1 by definition, with lower scores denoting a more favorable profile.
Physical activity and sedentariness | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  The International Physical Activity Questionnaire (IPAQ) will be used to evaluate the current physical activity level of the participants. The survey validity and reliability studies have been conducted in Turkey by Ozturk. The survey consists of 27 questions and 5 parts. Minimum value = 0 min/day of physical activity // Maximum value = 1440 min/day of physical activity. Higher scores imply a more physically active pattern.
  Objectively physical activity will be assessed by accelerometry
Dietary habits | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  A food frequency questionnaire (FFQ) conducted by a trained nutritionist. Based on dietary data from the FFQ, the investigators will calculate the Mediterranean Diet Score. Minimum value: 0 // Maximum value: 14. Higher scores mean a better outcome.
  PREDIMED adherence to the Mediterranean diet questionnaire will also be conducted by a trained nutritionist.
Others unhealthy habits | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  A seven-day self-reported tobacco and alcohol consumption logs will be used to determine smoking and alcohol intake registering total number of cigarettes and alcoholic units/day, time and situation in which both are consumed and cigarette type of alcoholic drink.
Nicotine dependence | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  The Fagerström Test for Nicotine Dependence will be used to measure patients' nicotine dependence. Minimum value: 0 // Maximum value: 10. Higher scores mean a worse outcome.
Sleep quality | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  Sleep quality will be determined by the Pittsburgh Sleep Quality Index (PSQI) scale. PSQI global score ranges from 0 to 21, with a score higher than 5 indicating poor sleep quality Objectively sleep quality will be assessed by accelerometry
Fecal microbiota analysis | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  A fecal sample (50-60 g) will be obtained and analyzed.
Molecular Characterization of Colon Tumor Tissue | Day of surgery
  Colon tumor tissue samples will be collected during surgical resection and analyzed using molecular techniques (e.g., gene expression profiling) to assess markers associated with tumor progression.
Cost-effectiveness analysis | At the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  We will calculate the ratio of incremental costs and incremental clinical benefits as the additional expenditure required to generate an additional unit of benefit, expressed as cost per quality-adjusted life-year (QALY) added, and calculated as CE = (Cost2-Cost1)/(QALY2-QALY1). EuroQol 5-dimension 5-level (EQ-5D-5L) will be used for QALY estimation. With regard to the cost measurements, we will follow the WHO recommendations for estimating costs contemplated in its CEA guidelines such as the cost of providing the intervention and costs of accessing the intervention.
Heart rate variability | Baseline (week 0), at preoperative conditions (week 5), at the end of the PPP intervention (week 17) and 1-year post-surgery (week 57).
  Participants will be lying in a supine position on a stretcher while the R-R signal will be assessed for 15 min (after 10 min of acclimation) using the Polar Ignite 2

CONTACTS AND LOCATIONS:
Overall Officials: Francisco J Amaro-Gahete, PhD, MD, Principal Investigator — Universidad de Granada
Locations (1):
- Department of Medical Physiology, Faculty of Medicine, University of Granada, Granada, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Bull FC, Al-Ansari SS, Biddle S, Borodulin K, Buman MP, Cardon G, Carty C, Chaput JP, Chastin S, Chou R, Dempsey PC, DiPietro L, Ekelund U, Firth J, Friedenreich CM, Garcia L, Gichu M, Jago R, Katzmarzyk PT, Lambert E, Leitzmann M, Milton K, Ortega FB, Ranasinghe C, Stamatakis E, Tiedemann A, Troiano RP, van der Ploeg HP, Wari V, Willumsen JF. World Health Organization 2020 guidelines on physical activity and sedentary behaviour. Br J Sports Med. 2020 Dec;54(24):1451-1462. doi: 10.1136/bjsports-2020-102955. PMID 33239350
- [Background] Mentella MC, Scaldaferri F, Ricci C, Gasbarrini A, Miggiano GAD. Cancer and Mediterranean Diet: A Review. Nutrients. 2019 Sep 2;11(9):2059. doi: 10.3390/nu11092059. PMID 31480794
- [Background] Cheville AL, Mustian K, Winters-Stone K, Zucker DS, Gamble GL, Alfano CM. Cancer Rehabilitation: An Overview of Current Need, Delivery Models, and Levels of Care. Phys Med Rehabil Clin N Am. 2017 Feb;28(1):1-17. doi: 10.1016/j.pmr.2016.08.001. PMID 27912990
- [Background] Carli F, Bousquet-Dion G, Awasthi R, Elsherbini N, Liberman S, Boutros M, Stein B, Charlebois P, Ghitulescu G, Morin N, Jagoe T, Scheede-Bergdahl C, Minnella EM, Fiore JF Jr. Effect of Multimodal Prehabilitation vs Postoperative Rehabilitation on 30-Day Postoperative Complications for Frail Patients Undergoing Resection of Colorectal Cancer: A Randomized Clinical Trial. JAMA Surg. 2020 Mar 1;155(3):233-242. doi: 10.1001/jamasurg.2019.5474. PMID 31968063
- [Background] Fulop A, Lakatos L, Susztak N, Szijarto A, Banky B. The effect of trimodal prehabilitation on the physical and psychological health of patients undergoing colorectal surgery: a randomised clinical trial. Anaesthesia. 2021 Jan;76(1):82-90. doi: 10.1111/anae.15215. Epub 2020 Aug 6. PMID 32761611
- [Background] Minnella EM, Bousquet-Dion G, Awasthi R, Scheede-Bergdahl C, Carli F. Multimodal prehabilitation improves functional capacity before and after colorectal surgery for cancer: a five-year research experience. Acta Oncol. 2017 Feb;56(2):295-300. doi: 10.1080/0284186X.2016.1268268. Epub 2017 Jan 12. PMID 28079430
- [Background] Frawley HC, Lin KY, Granger CL, Higgins R, Butler M, Denehy L. An allied health rehabilitation program for patients following surgery for abdomino-pelvic cancer: a feasibility and pilot clinical study. Support Care Cancer. 2020 Mar;28(3):1335-1350. doi: 10.1007/s00520-019-04931-w. Epub 2019 Jun 27. PMID 31250182
- [Background] Slankamenac K, Graf R, Barkun J, Puhan MA, Clavien PA. The comprehensive complication index: a novel continuous scale to measure surgical morbidity. Ann Surg. 2013 Jul;258(1):1-7. doi: 10.1097/SLA.0b013e318296c732. PMID 23728278
- [Background] Slankamenac K, Nederlof N, Pessaux P, de Jonge J, Wijnhoven BP, Breitenstein S, Oberkofler CE, Graf R, Puhan MA, Clavien PA. The comprehensive complication index: a novel and more sensitive endpoint for assessing outcome and reducing sample size in randomized controlled trials. Ann Surg. 2014 Nov;260(5):757-62; discussion 762-3. doi: 10.1097/SLA.0000000000000948. PMID 25379846

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-06-11): https://cdn.clinicaltrials.gov/large-docs/05/NCT05379205/SAP_000.pdf